CLINICAL TRIAL: NCT00443261
Title: Phase I Study of Azacitidine in Combination With Cisplatin Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Azacitidine and Cisplatin for Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual problems
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10498
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Squamous Cell Carcinoma
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Azacitidine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (SCCHN) (Experimental): Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck Patients will receive Azacitidine and cisplatin.
  Interventions: Drug: Azacitidine; Drug: Cisplatin

INTERVENTIONS:
Drug: Azacitidine — SC azacitidine
  Other Names: 5-azacitidine, Vidaza
Drug: Cisplatin — cisplatin 75 mg/m^2 day 8 every 28 days
  Other Names: cis-platinum, platinol

SUMMARY:
To evaluate the safety and toxicity of azacitidine (5-azacitidine, Vidaza®) and cisplatin combination in patients with squamous cell carcinoma of head and neck (SCCHN).

DETAILED DESCRIPTION:
Open-label, non-randomized and dose escalation study in which groups of 3-6 patients with squamous cell carcinoma of the head and neck will receive sequentially increased dosages of azacitidine SC injection in combination with a fixed dose of cisplatin IV injection until dose-limiting toxicity is demonstrated in 2 of the 6 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven SCCHN that is either metastatic or has persisted or recurred following definitive surgery and/or radiation therapy, and is not amenable to salvage surgical resection.
* Patients may have received previous chemotherapy and/or biological treatment (such as cetuximab) for the recurrent or metastatic disease. Prior treatment must have been completed at least 28 days (42 days for nitrosoureas or mitomycin C) prior to entering the study and all toxicities must have been resolved.
* Prior radiation must have been completed at least 28 days before entry into the study and all toxicities must have been resolved (no more than 3000 cGy to fields including substantial marrow).
* Surgery must have been completed at least 28 days before entry into the study and all complications/adverse events must have been resolved.
* Patients must have at least one lesion amenable to serial biopsy.
* Age greater than 18 years.
* ECOG performance status less than 2 (Karnofsky greater than 60%).
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function
* Patients must not be planning to receive any other concurrent therapy (ie, radiation, chemotherapy, immunotherapy, biological therapy or gene therapy) for SCCHN while they are on this study.
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine treatment.

Exclusion Criteria:

* Patients must not be planning to receive any other concurrent therapy (ie, radiation, chemotherapy, immunotherapy, biological therapy, investigational agents or gene therapy) for SCCHN while they are on this study.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to azacitidine, cisplatin and mannitol or other agents used in study.
* Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients known to be HIV-positive are not eligible because of the potential to confound this study's endpoints.
* No prior malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease-free for five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K. Williamson, MD, Study Director — University of Kansas Medical Center; Chao H. Huang, MD, Study Chair — University of Kansas Medical Center
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: SCCHN: Intervention:
  Azacitidine: SC daily X 5 every 28 days azacitidine at assigned dose ranging from 37 to 110 mg/M^2/day.
  Cisplatin: cisplatin 75 mg/m^2 day 8 every 28 days
Period: Overall Study
Arm/Group | Arm 1: SCCHN
Started | 1
Accrual in 10 Months | 1 (Patient died due to progressive disease after cycle 1 of treatment)
Completed | 0 (Study terminated due to poor accrual and only patient enrolled died)
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- 1: SCCHN: Azacitidine and cisplatin
  Azacitidine: SC azacitidine
  Cisplatin: cisplatin 75 mg/m2 day 8 every 28 days
Arm/Group | 1: SCCHN
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 52 (0)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety and Toxicity of Azacitidine (5-azacytidine, Vidaza®) and Cisplatin Combination
Description: Although response is not the primary endpoint of this trial, patients with measurable disease will by assessed by standard criteria. For the purpose of this study, patients should be re-evaluated every 8 weeks by imaging study. In addition to baseline scan, confirmatory scans will also be obtained 4 weeks following initial documentation of an objective response.
Time Frame: Weeks 1-12, 24, 36
Population: The 1 patient enrolled in the study died after cycle 1 with rapidly progressing cancer. Therefore, no data to analyze for primary outcome measure.
Groups:
- Arm 1: SCCHN: Azacitidine and cisplatin
  Azacitidine: SC azacitidine
  Cisplatin: cisplatin 75 mg/m^2 day 8 every 28 days
Arm/Group | Arm 1: SCCHN
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | 1: SCCHN
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: SCCHN (N=1)
Pnemonia (Infections and infestations) | 1 (1) — Patient admitted 10 days after treatment with pneumonia secondary to rapidly progressive cancer. She died 6/27/07

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No